CLINICAL TRIAL: NCT00469300
Title: A Multicenter, Placebo Controlled, Randomized, Double Blind, Subject Initiated Study of the Safety and Efficacy of the Electrokinetic Transdermal System (ETS) With Acyclovir Gel for the Episodic Treatment of Herpes Labialis
Brief Title: Iontophoretic Application of Acyclovir Gel to Treat Cold Sores
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Transport Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPI-H-221
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2008-02-04 (Estimated); Status verified 2008-01

CONDITIONS: Herpes Labialis
Keywords: herpes labialis; cold sore; acyclovir; iontophoresis; topical
MeSH Terms: conditions — Herpes Labialis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Iontophoretic delivery of acyclovir

SUMMARY:
Currently approved drugs for the treatment of herpes labialis (cold sores) exhibit low levels of efficacy due to the limited ability of the drugs to penetrate the skin to the sites where the herpes virus is replicating. Iontophoresis uses electric current to enhance delivery of drugs through the skin. This trial is testing a new iontophoretic device with a new acyclovir gel to treat cold sores.

DETAILED DESCRIPTION:
This is a multicenter, placebo controlled, randomized, double blind, subject initiated study of the safety and efficacy of a single, 10-minute, topical iontophoretic application of a novel acyclovir 5% gel for the episodic treatment of recurrent herpes labialis. The design of the trial will also allow the comparison of the efficacy of a single iontophoretic treatment with acyclovir gel within 1 hour of first signs and/or symptoms of a herpetic episode to the efficacy of a single iontophoretic treatment with acyclovir gel 6 to18 hours after first signs and/or symptoms. Approximately 810 subjects will be enrolled to treat about 80 subjects in each of three treatment arms. Depending upon how the subject has been randomized into the trial, the subject will receive either: 1) an iontophoretic treatment with active gel within 1 hour of first signs/and or symptoms, followed 6-18 hours later by a second treatment with placebo gel; 2) an iontophoretic treatment with placebo gel within 1 hour of first signs/and or symptoms, followed 6-18 hours later by a second treatment with active gel; or 3) an iontophoretic treatment with placebo gel within 1 hour of first signs/and or symptoms, followed 6-18 hours later by a second treatment with placebo gel. After being enrolled and randomized into the study, subjects will be sent home with a locked kit containing the iontophoretic device with either active or placebo gel. At first signs and/or symptoms of a recurrent herpetic episode (prodromal or erythema), the lesion will be confirmed by telephone interview with the subject and, upon confirmation of the lesion, the subject will be given the combination to the locked kit and instructed to begin treatment immediately. The subject will then be instructed to return to the clinic within 6 to 18 hours of first signs and/or symptoms for a second iontophoretic treatment, appropriate to the treatment arm into which they have been randomized, and an evaluation. The subject will visit the clinic for daily follow-up evaluations for 3 to 14 days following the first treatment and will be called 2 weeks after their last clinic visit for a final safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject 18-75 years of age
2. Female subjects must be using a medically acceptable form of birth control during the study.
3. Subject must have a history of recurrent herpes labialis and report at least 3 recurrences during the preceding 12 months.
4. Subject must provide voluntary written informed consent to participate in this study.

Exclusion Criteria:

1. Subjects with a pacemaker, a history of cardiac arrhythmias or conduction abnormalities.
2. Any evidence of active malignancy or immunodeficient disease within the last 30 days. Subjects who have completed therapy and are considered unlikely to relapse or who have had surgery and do not have any evidence of disease, are eligible for the study.
3. Subject requires chronic use of immunomodifying drugs (e.g. systemic steroids) or topical steroids on or near the face; use of inhaled steroids does not exclude a subject from the study.
4. Subject requires chronic use of anti-viral medication.
5. History of allergic or adverse response to acyclovir, or any related anti-viral drug, or the gel base.
6. In females of childbearing potential, a positive urine pregnancy test at time of screening.
7. Nursing mothers.
8. Subjects with an implantable electronic device.
9. Subject has any body piercing in or around the area ordinarily affected by cold sores.
10. Subject is considered unreliable or unable to understand or follow the protocol directions or is unable to comprehend or satisfactorily assess a herpetic lesion as determined by Investigator or designee at screening.
11. Subject has abnormal skin conditions (e.g. acne, eczema, psoriasis, albinism, or chronic vesiculobullous disorders) that occur in the area ordinarily affected by cold sores or has significant facial hair in the area of the cold sore that might affect the normal course of the cold sore or might impair accurate evaluation of the cold sore lesion.
12. Subject has had an infection with HSV-1 isolates know to be resistant to acyclovir, valacyclovir, famciclovir, or ganciclovir.
13. Subject has had a herpes vaccine.
14. Subject is currently enrolled in another clinical trial involving the use of a drug and/or a device.
15. Subject has previously participated in the current study (TPI-H-221).
16. Subject requires chronic use of analgesics, pain medication or non-steroidal anti-inflammatory agents (NSAIDs).
17. Subject has a recent history of renal dysfunction or serious hepatic disease.
18. Subject has a history of alcoholism or drug abuse within the preceding 12 months.
19. Subject shares a household with another subject already enrolled in the study (TPI-H-221). If the other household member has already completed the study, then the currently enrolling subject is not excluded.
20. Subject is institutionalized.
21. Any history which, in the Investigator's judgment, makes the subject ineligible or places the subject at undue risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Estimated)
Dates: Start 2007-04; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Clinician assessed duration of the herpetic episode measured from the time of treatment until the lesion is healed. | Lesion assessments for a minimum of 3 consecutive days and a maximum of 14 days.

SECONDARY OUTCOMES:
Clinician assessed: Prevention of progression to a classical lesion;Duration of classical herpetic lesions; Duration of herpetic lesions; Duration of the herpetic lesion hard scab; Duration until complete healing of the herpetic episode; | Lesion assessment for a minimum of 3 consecutive days and a maximum of 14 consecutive days.

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Morrel, PhD, Study Director — Transport Pharmaceuticals, Inc.
Locations (13):
- United States (13):
  - Radiant Research Birmingham, Birmingham, Alabama
  - Radiant Research Santa Rosa, Santa Rosa, California
  - Radiant Research St. Petersburg, Pinellas Park, Florida
  - Radiant Research Chicago, Chicago, Illinois
  - Radiant Research Minneapolis, Edina, Minnesota
  - Radiant Research St. Louis, St Louis, Missouri
  - Rochester Clinical Research, Inc., Rochester, New York
  - Radiant Research Cincinnati, Cincinnati, Ohio
  - Radiant Research Akron, Mogadore, Ohio
  - OMEGA Medical Research, Warwick, Rhode Island
  - Radiant Research Greer, Greer, South Carolina
  - Radiant Research Dallas North, Dallas, Texas
  - Radiant Research San Antonio, San Antonio, Texas

REFERENCES:
- [Background] Morrel EM, Spruance SL, Goldberg DI; Iontophoretic Acyclovir Cold Sore Study Group. Topical iontophoretic administration of acyclovir for the episodic treatment of herpes labialis: a randomized, double-blind, placebo-controlled, clinic-initiated trial. Clin Infect Dis. 2006 Aug 15;43(4):460-7. doi: 10.1086/505872. Epub 2006 Jul 3. PMID 16838235
- See also: Mayo Clinic Cold Sore Information — http://www.mayoclinic.com/invoke.cfm?id=DS00358